CLINICAL TRIAL: NCT05307965
Title: Stent Retriever Thrombectomy for Thrombus Burden Reduction in Patients With Acute Myocardial Infarction - RETRIEVE-AMI Study
Brief Title: RETRIEVE-AMI Study
Acronym: RETRIEVE-AMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Oxford University Hospitals NHS Trust (Other)
Collaborators: Medtronic (Industry); Terumo Corporation (Industry)
Responsible Party: Principal Investigator, Giovanni Luigi De Maria, Primary Investigator, Oxford University Hospitals NHS Trust
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15488
Record Dates: First submitted 2022-03-02; First posted 2022-04-01 (Actual); Results first posted 2025-09-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: Myocardial Infarction; Thrombus; Coronary Artery Disease
Keywords: Myocardial Infarction; Percutaneous coronary intervention; Stent Retriever; Thrombus Aspiration
MeSH Terms: conditions — Myocardial Infarction; Thrombosis; Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Intervention Model Description: The study will consist of 3 arms. Eligible participants will be 1:1:1 randomised to receive either standalone percutaneous coronary intervention (PCI) (Arm 1), thrombus aspiration + PCI (Arm 2) or retriever thrombectomy + PCI (Arm 3).
Who Masked: Outcomes Assessor
Masking Description: Due to the interventional nature of the trial, masking is not feasible for operators, the clinical care team and participants. However, analysis of the OCT-derived primary and secondary end-points will be conducted offline in a blinded fashion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standalone Percutaneous Coronary Intervention (Active Comparator): Participants will have standard of care treatment. They will undergo PCI with devices and techniques driven by clinical decision making at the patient level and institutional level, and carried out in accordance with the Oxford University Hospitals NHS Foundation Trust department guidelines.
  Interventions: Procedure: Percutaneous Coronary Intervention
- Percutaneous Coronary Intervention and Thrombus Aspiration (Active Comparator): Participants will have standard of care treatment with manual thrombectomy catheter and PCI. They will undergo PCI with devices and techniques driven by clinical decision making at the patient level and institutional level, and carried out in accordance with the Oxford University Hospitals NHS Foundation Trust department guidelines.
  Interventions: Procedure: Percutaneous Coronary Intervention; Procedure: Thrombus Aspiration
- Percutaneous Coronary Intervention and Retriever Thrombectomy (Experimental): Participants randomised to the stent-retriever thrombectomy arm of the RETRIEVE AMI trial will undergo stent-retriever thrombectomy with the SolitaireTM X Revascularisation Device.
  Interventions: Device: Retriever Thrombectomy; Procedure: Percutaneous Coronary Intervention

INTERVENTIONS:
Device: Retriever Thrombectomy — The SolitaireTM X revascularisation device is a self-expanding stent designed for dynamic clot integration with radiopaque markers that enhance visualisation of the optimal working length. After a thrombotic occlusion has been identified and crossed with a guidewire, the stent-retriever thrombectomy proceeds. A microcatheter (e.g., PhenomTM, MarksmanTM) is advanced over the guidewire and once it has traversed the thrombotic occlusion, the SolitaireTM X device is advanced through the microcatheter until the usable length of the stent extends past each side of the thrombus in the vessel. As the microcatheter is retracted to the proximal radiopaque marker of the stent, the stent self-expands and entangles the thrombus. The microcatheter and SolitaireTM X Revascularisation Device are withdrawn as a unit into the guide catheter under continuous aspiration. PCI then proceeds driven by clinical decision making and department guidelines.
  Other Names: SolitaireTM X Revascularisation Device; Stent Retriever
  Arms: Percutaneous Coronary Intervention and Retriever Thrombectomy
Procedure: Percutaneous Coronary Intervention — Standard of care
Procedure: Thrombus Aspiration — Standard of care treatment with manual thrombectomy catheter
  Other Names: Aspiration-assisted thrombectomy
  Arms: Percutaneous Coronary Intervention and Thrombus Aspiration

SUMMARY:
Heart attacks are caused by the sudden formation of a clot inside a diseased coronary artery which reduces blood flow beyond the blockage site. During conventional treatment of the blockage with what is known as a stent; a stainless steel tub that keeps the artery open, the clot that has formed is disrupted and is pushed further down leading to damage in smaller blood vessels supplying the heart muscle. This additional damage can lead to long-term heart muscle damage influencing recovery and wellbeing. The original concept that was tested to prevent this 'clot shower' was that of a suction device to withdraw the clot before stenting. However, this approach has not translated to patient benefit. Amongst the reasons put forward for the inefficacy of the suction device was that it does not remove the entire clot as it does not interact with it. A new device that physically interacts with the clot and traps it before pulling it out - the stent retriever - is now routinely used in stroke therapy to remove clots in the arteries supplying the brain. This device has been successfully used as a last resort to remove clots in a small number of heart attacks. The investigators hypothesize that stent retriever therapy will be more effective in clot removal than the current standard of care; suction or stenting. To study this, the investigators propose the RETRIEVE-AMI randomised controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Primary PCI patient with ST elevation myocardial infarction (STEMI)
* TIMI 0/1 flow at presentation
* Angiographic thrombus score ≥ 4
* Vessel diameter at site of occlusion ≥ 3.0 mm (measured by quantitative coronary angiography)

Exclusion Criteria:

* Female participant who is pregnant or lactating
* Participant with known hypersensitivity to nickel-titanium
* Unconscious at presentation
* Late presenter (pain to wire time > 12 h)
* Class Killip III/IV and/or profound bradycardia (Heart rate < 40 bpm)
* Known history of kidney failure
* Ostial occlusion
* Highly tortuous vessel
* Highly calcified vessel
* Suspected (angiographically) spontaneous coronary artery dissection
* Stent thrombosis
* Previous stent implanted proximal to the occlusion site
* Previous coronary artery bypass graft surgery (CABG)
* Previous STEMI/Transient Ischemic Attack/Stroke
* Known anaemia (Hemoglobin <9)

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2022-05-06 (Actual); Primary Completion 2024-10-24 (Actual); Study Completion 2025-05-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Luigi De Maria, Principal Investigator — Oxford University Hospitals NHS Trust
Locations (1):
- Oxford Heart Centre, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: No
There is no plan to make IPD available to other researchers unless requested and upon the discretion of the Chief Investigator

REFERENCES:
- [Background] Nowbar AN, Gitto M, Howard JP, Francis DP, Al-Lamee R. Mortality From Ischemic Heart Disease. Circ Cardiovasc Qual Outcomes. 2019 Jun;12(6):e005375. doi: 10.1161/CIRCOUTCOMES.118.005375. Epub 2019 Jun 4. PMID 31163980
- [Background] Braunwald E. The treatment of acute myocardial infarction: the Past, the Present, and the Future. Eur Heart J Acute Cardiovasc Care. 2012 Apr;1(1):9-12. doi: 10.1177/2048872612438026. PMID 24062883
- [Background] Niccoli G, Scalone G, Lerman A, Crea F. Coronary microvascular obstruction in acute myocardial infarction. Eur Heart J. 2016 Apr 1;37(13):1024-33. doi: 10.1093/eurheartj/ehv484. Epub 2015 Sep 12. PMID 26364289
- [Background] De Maria GL, Patel N, Wolfrum M, Fahrni G, Kassimis G, Porto I, Dawkins S, Choudhury RP, Forfar JC, Prendergast BD, Channon KM, Kharbanda RK, Garcia-Garcia HM, Banning AP. The influence of coronary plaque morphology assessed by optical coherence tomography on final microvascular function after stenting in patients with ST-elevation myocardial infarction. Coron Artery Dis. 2017 May;28(3):198-208. doi: 10.1097/MCA.0000000000000458. PMID 27926579
- [Background] Vlaar PJ, Svilaas T, van der Horst IC, Diercks GF, Fokkema ML, de Smet BJ, van den Heuvel AF, Anthonio RL, Jessurun GA, Tan ES, Suurmeijer AJ, Zijlstra F. Cardiac death and reinfarction after 1 year in the Thrombus Aspiration during Percutaneous coronary intervention in Acute myocardial infarction Study (TAPAS): a 1-year follow-up study. Lancet. 2008 Jun 7;371(9628):1915-20. doi: 10.1016/S0140-6736(08)60833-8. PMID 18539223
- [Background] Jolly SS, Cairns JA, Yusuf S, Rokoss MJ, Gao P, Meeks B, Kedev S, Stankovic G, Moreno R, Gershlick A, Chowdhary S, Lavi S, Niemela K, Bernat I, Cantor WJ, Cheema AN, Steg PG, Welsh RC, Sheth T, Bertrand OF, Avezum A, Bhindi R, Natarajan MK, Horak D, Leung RC, Kassam S, Rao SV, El-Omar M, Mehta SR, Velianou JL, Pancholy S, Dzavik V; TOTAL Investigators. Outcomes after thrombus aspiration for ST elevation myocardial infarction: 1-year follow-up of the prospective randomised TOTAL trial. Lancet. 2016 Jan 9;387(10014):127-35. doi: 10.1016/S0140-6736(15)00448-1. Epub 2015 Oct 22. PMID 26474811
- [Background] Lagerqvist B, Frobert O, Olivecrona GK, Gudnason T, Maeng M, Alstrom P, Andersson J, Calais F, Carlsson J, Collste O, Gotberg M, Hardhammar P, Ioanes D, Kallryd A, Linder R, Lundin A, Odenstedt J, Omerovic E, Puskar V, Todt T, Zelleroth E, Ostlund O, James SK. Outcomes 1 year after thrombus aspiration for myocardial infarction. N Engl J Med. 2014 Sep 18;371(12):1111-20. doi: 10.1056/NEJMoa1405707. Epub 2014 Sep 1. PMID 25176395
- [Background] Higuma T, Soeda T, Yamada M, Yokota T, Yokoyama H, Izumiyama K, Nishizaki F, Minami Y, Xing L, Yamamoto E, Lee H, Okumura K, Jang IK. Does Residual Thrombus After Aspiration Thrombectomy Affect the Outcome of Primary PCI in Patients With ST-Segment Elevation Myocardial Infarction?: An Optical Coherence Tomography Study. JACC Cardiovasc Interv. 2016 Oct 10;9(19):2002-2011. doi: 10.1016/j.jcin.2016.06.050. PMID 27712735
- [Background] Bhindi R, Kajander OA, Jolly SS, Kassam S, Lavi S, Niemela K, Fung A, Cheema AN, Meeks B, Alexopoulos D, Kocka V, Cantor WJ, Kaivosoja TP, Shestakovska O, Gao P, Stankovic G, Dzavik V, Sheth T. Culprit lesion thrombus burden after manual thrombectomy or percutaneous coronary intervention-alone in ST-segment elevation myocardial infarction: the optical coherence tomography sub-study of the TOTAL (ThrOmbecTomy versus PCI ALone) trial. Eur Heart J. 2015 Aug 1;36(29):1892-900. doi: 10.1093/eurheartj/ehv176. Epub 2015 May 20. PMID 25994742
- [Background] Berkhemer OA, Fransen PS, Beumer D, van den Berg LA, Lingsma HF, Yoo AJ, Schonewille WJ, Vos JA, Nederkoorn PJ, Wermer MJ, van Walderveen MA, Staals J, Hofmeijer J, van Oostayen JA, Lycklama a Nijeholt GJ, Boiten J, Brouwer PA, Emmer BJ, de Bruijn SF, van Dijk LC, Kappelle LJ, Lo RH, van Dijk EJ, de Vries J, de Kort PL, van Rooij WJ, van den Berg JS, van Hasselt BA, Aerden LA, Dallinga RJ, Visser MC, Bot JC, Vroomen PC, Eshghi O, Schreuder TH, Heijboer RJ, Keizer K, Tielbeek AV, den Hertog HM, Gerrits DG, van den Berg-Vos RM, Karas GB, Steyerberg EW, Flach HZ, Marquering HA, Sprengers ME, Jenniskens SF, Beenen LF, van den Berg R, Koudstaal PJ, van Zwam WH, Roos YB, van der Lugt A, van Oostenbrugge RJ, Majoie CB, Dippel DW; MR CLEAN Investigators. A randomized trial of intraarterial treatment for acute ischemic stroke. N Engl J Med. 2015 Jan 1;372(1):11-20. doi: 10.1056/NEJMoa1411587. Epub 2014 Dec 17. PMID 25517348
- [Background] Goyal M, Demchuk AM, Menon BK, Eesa M, Rempel JL, Thornton J, Roy D, Jovin TG, Willinsky RA, Sapkota BL, Dowlatshahi D, Frei DF, Kamal NR, Montanera WJ, Poppe AY, Ryckborst KJ, Silver FL, Shuaib A, Tampieri D, Williams D, Bang OY, Baxter BW, Burns PA, Choe H, Heo JH, Holmstedt CA, Jankowitz B, Kelly M, Linares G, Mandzia JL, Shankar J, Sohn SI, Swartz RH, Barber PA, Coutts SB, Smith EE, Morrish WF, Weill A, Subramaniam S, Mitha AP, Wong JH, Lowerison MW, Sajobi TT, Hill MD; ESCAPE Trial Investigators. Randomized assessment of rapid endovascular treatment of ischemic stroke. N Engl J Med. 2015 Mar 12;372(11):1019-30. doi: 10.1056/NEJMoa1414905. Epub 2015 Feb 11. PMID 25671798
- [Background] Campbell BC, Mitchell PJ, Kleinig TJ, Dewey HM, Churilov L, Yassi N, Yan B, Dowling RJ, Parsons MW, Oxley TJ, Wu TY, Brooks M, Simpson MA, Miteff F, Levi CR, Krause M, Harrington TJ, Faulder KC, Steinfort BS, Priglinger M, Ang T, Scroop R, Barber PA, McGuinness B, Wijeratne T, Phan TG, Chong W, Chandra RV, Bladin CF, Badve M, Rice H, de Villiers L, Ma H, Desmond PM, Donnan GA, Davis SM; EXTEND-IA Investigators. Endovascular therapy for ischemic stroke with perfusion-imaging selection. N Engl J Med. 2015 Mar 12;372(11):1009-18. doi: 10.1056/NEJMoa1414792. Epub 2015 Feb 11. PMID 25671797
- [Background] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510
- [Background] Saver JL, Goyal M, Bonafe A, Diener HC, Levy EI, Pereira VM, Albers GW, Cognard C, Cohen DJ, Hacke W, Jansen O, Jovin TG, Mattle HP, Nogueira RG, Siddiqui AH, Yavagal DR, Baxter BW, Devlin TG, Lopes DK, Reddy VK, du Mesnil de Rochemont R, Singer OC, Jahan R; SWIFT PRIME Investigators. Stent-retriever thrombectomy after intravenous t-PA vs. t-PA alone in stroke. N Engl J Med. 2015 Jun 11;372(24):2285-95. doi: 10.1056/NEJMoa1415061. Epub 2015 Apr 17. PMID 25882376
- [Background] Bhoopalan K, Rajendran R, Alagarsamy S, Kesavamoorthy N. Successful extraction of refractory thrombus from an ectatic coronary artery using stent retriever during primary angioplasty for acute myocardial infarction: a case report. Eur Heart J Case Rep. 2019 Jan 9;3(1):yty161. doi: 10.1093/ehjcr/yty161. eCollection 2019 Mar. PMID 31020237
- [Background] Patel N, Badiye A, Yavagal DR, Mendoza CE. Stent-Based Mechanical Thrombectomy in Left Main Coronary Artery Thrombus Presenting as ST-Segment Elevation Myocardial Infarction. JACC Cardiovasc Interv. 2017 Feb 13;10(3):302-303. doi: 10.1016/j.jcin.2016.10.038. Epub 2017 Jan 18. No abstract available. PMID 28109870
- [Background] Kajander OA, Koistinen LS, Eskola M, Huhtala H, Bhindi R, Niemela K, Jolly SS, Sheth T; TOTAL-OCT Substudy Investigators. Feasibility and repeatability of optical coherence tomography measurements of pre-stent thrombus burden in patients with STEMI treated with primary PCI. Eur Heart J Cardiovasc Imaging. 2015 Jan;16(1):96-107. doi: 10.1093/ehjci/jeu175. Epub 2014 Sep 19. PMID 25240168
- [Background] Ali ZA, Karimi Galougahi K, Maehara A, Shlofmitz RA, Ben-Yehuda O, Mintz GS, Stone GW. Intracoronary Optical Coherence Tomography 2018: Current Status and Future Directions. JACC Cardiovasc Interv. 2017 Dec 26;10(24):2473-2487. doi: 10.1016/j.jcin.2017.09.042. PMID 29268880
- [Background] De Maria GL, Alkhalil M, Wolfrum M, Fahrni G, Borlotti A, Gaughran L, Dawkins S, Langrish JP, Lucking AJ, Choudhury RP, Porto I, Crea F, Dall'Armellina E, Channon KM, Kharbanda RK, Banning AP. Index of Microcirculatory Resistance as a Tool to Characterize Microvascular Obstruction and to Predict Infarct Size Regression in Patients With STEMI Undergoing Primary PCI. JACC Cardiovasc Imaging. 2019 May;12(5):837-848. doi: 10.1016/j.jcmg.2018.02.018. Epub 2018 Apr 18. PMID 29680355
- [Background] Tu S, Barbato E, Koszegi Z, Yang J, Sun Z, Holm NR, Tar B, Li Y, Rusinaru D, Wijns W, Reiber JH. Fractional flow reserve calculation from 3-dimensional quantitative coronary angiography and TIMI frame count: a fast computer model to quantify the functional significance of moderately obstructed coronary arteries. JACC Cardiovasc Interv. 2014 Jul;7(7):768-77. doi: 10.1016/j.jcin.2014.03.004. PMID 25060020
- [Background] Tu S, Xu L, Ligthart J, Xu B, Witberg K, Sun Z, Koning G, Reiber JH, Regar E. In vivo comparison of arterial lumen dimensions assessed by co-registered three-dimensional (3D) quantitative coronary angiography, intravascular ultrasound and optical coherence tomography. Int J Cardiovasc Imaging. 2012 Aug;28(6):1315-27. doi: 10.1007/s10554-012-0016-6. Epub 2012 Jan 20. PMID 22261998
- [Background] Albers GW, Marks MP, Kemp S, Christensen S, Tsai JP, Ortega-Gutierrez S, McTaggart RA, Torbey MT, Kim-Tenser M, Leslie-Mazwi T, Sarraj A, Kasner SE, Ansari SA, Yeatts SD, Hamilton S, Mlynash M, Heit JJ, Zaharchuk G, Kim S, Carrozzella J, Palesch YY, Demchuk AM, Bammer R, Lavori PW, Broderick JP, Lansberg MG; DEFUSE 3 Investigators. Thrombectomy for Stroke at 6 to 16 Hours with Selection by Perfusion Imaging. N Engl J Med. 2018 Feb 22;378(8):708-718. doi: 10.1056/NEJMoa1713973. Epub 2018 Jan 24. PMID 29364767
- [Background] Tarasow E, Abdulwahed Saleh Ali A, Lewszuk A, Walecki J. Measurements of the middle cerebral artery in digital subtraction angiography and MR angiography. Med Sci Monit. 2007 May;13 Suppl 1:65-72. PMID 17507888
- [Background] Saver JL, Jahan R, Levy EI, Jovin TG, Baxter B, Nogueira RG, Clark W, Budzik R, Zaidat OO; SWIFT Trialists. Solitaire flow restoration device versus the Merci Retriever in patients with acute ischaemic stroke (SWIFT): a randomised, parallel-group, non-inferiority trial. Lancet. 2012 Oct 6;380(9849):1241-9. doi: 10.1016/S0140-6736(12)61384-1. Epub 2012 Aug 26. PMID 22932715
- [Background] Kinnaird T, Kwok CS, Davies R, Calvert PA, Anderson R, Gallagher S, Sirker A, Ludman P, deBelder M, Stables R, Johnson TW, Kontopantelis E, Curzen N, Mamas M; British Cardiovascular Intervention Society and the National Institute for Cardiovascular Outcomes Research. Coronary perforation complicating percutaneous coronary intervention in patients presenting with an acute coronary syndrome: An analysis of 1013 perforation cases from the British Cardiovascular Intervention Society database. Int J Cardiol. 2020 Jan 15;299:37-42. doi: 10.1016/j.ijcard.2019.06.034. Epub 2019 Jun 14. PMID 31253528
- [Background] Kobayashi N, Mintz GS, Witzenbichler B, Metzger DC, Rinaldi MJ, Duffy PL, Weisz G, Stuckey TD, Brodie BR, Parvataneni R, Kirtane AJ, Stone GW, Maehara A. Prevalence, Features, and Prognostic Importance of Edge Dissection After Drug-Eluting Stent Implantation: An ADAPT-DES Intravascular Ultrasound Substudy. Circ Cardiovasc Interv. 2016 Jul;9(7):e003553. doi: 10.1161/CIRCINTERVENTIONS.115.003553. PMID 27402854
- [Background] Myint PK, Kwok CS, Roffe C, Kontopantelis E, Zaman A, Berry C, Ludman PF, de Belder MA, Mamas MA; British Cardiovascular Intervention Society and the National Institute for Cardiovascular Outcomes Research. Determinants and Outcomes of Stroke Following Percutaneous Coronary Intervention by Indication. Stroke. 2016 Jun;47(6):1500-7. doi: 10.1161/STROKEAHA.116.012700. Epub 2016 May 10. PMID 27165953
- [Background] Jolly SS, James S, Dzavik V, Cairns JA, Mahmoud KD, Zijlstra F, Yusuf S, Olivecrona GK, Renlund H, Gao P, Lagerqvist B, Alazzoni A, Kedev S, Stankovic G, Meeks B, Frobert O. Thrombus Aspiration in ST-Segment-Elevation Myocardial Infarction: An Individual Patient Meta-Analysis: Thrombectomy Trialists Collaboration. Circulation. 2017 Jan 10;135(2):143-152. doi: 10.1161/CIRCULATIONAHA.116.025371. Epub 2016 Dec 9. PMID 27941066
- [Background] Shoji S, Kohsaka S, Kumamaru H, Sawano M, Shiraishi Y, Ueda I, Noma S, Suzuki M, Numasawa Y, Hayashida K, Yuasa S, Miyata H, Fukuda K. Stroke After Percutaneous Coronary Intervention in the Era of Transradial Intervention. Circ Cardiovasc Interv. 2018 Dec;11(12):e006761. doi: 10.1161/CIRCINTERVENTIONS.118.006761. PMID 30545258
- [Background] Amabile N, Hammas S, Fradi S, Souteyrand G, Veugeois A, Belle L, Motreff P, Caussin C. Intra-coronary thrombus evolution during acute coronary syndrome: regression assessment by serial optical coherence tomography analyses. Eur Heart J Cardiovasc Imaging. 2015 Apr;16(4):433-40. doi: 10.1093/ehjci/jeu228. Epub 2014 Nov 26. PMID 25428947

RESULTS

PARTICIPANT FLOW:
Period: At Randomisation
Arm/Group | Standalone Percutaneous Coronary Intervention | Percutaneous Coronary Intervention and Thrombus Aspiration | Percutaneous Coronary Intervention and Retriever Thrombectomy
Started | 27 | 27 | 27
Completed | 27 | 26 | 27
Not Completed | 0 | 1 | 0
Period: Flow Following Randomisation
Arm/Group | Standalone Percutaneous Coronary Intervention | Percutaneous Coronary Intervention and Thrombus Aspiration | Percutaneous Coronary Intervention and Retriever Thrombectomy
Started | 28 | 27 | 26
Completed | 28 | 26 | 26
Not Completed | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standalone Percutaneous Coronary Intervention | Percutaneous Coronary Intervention and Thrombus Aspiration | Percutaneous Coronary Intervention and Retriever Thrombectomy | Total
Number analyzed (Participants) | 27 | 27 | 27 | 81
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (12) | 63 (12) | 63 (13) | 64 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 5 | 4 | 12
  Male | 24 | 22 | 23 | 69
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United Kingdom | 27 | 27 | 27 | 81

OUTCOME MEASURES:

1. Primary Outcome: Thrombus Volume (mm^3)
Description: Assessed with Optical Coherence Tomography [OCT]
Time Frame: During PCI prior to stent implantation (typically 30 min from start of procedure)
Population: The OCT run for one patient was not analysable due to slow flow precluding good blood clearance for a reliable measurement.
Measure: Median (Inter-Quartile Range); unit: mm^3
Arm/Group | Standalone Percutaneous Coronary Intervention | Percutaneous Coronary Intervention and Thrombus Aspiration | Percutaneous Coronary Intervention and Retriever Thrombectomy
Number analyzed (Participants) | 27 | 26 | 27
mm^3 | 9.8 [4.5 to 18.1] | 4.8 [1.8 to 8.4] | 7.7 [2.3 to 18.6]

2. Primary Outcome: Device-related Target Vessel Complications
Description: Assessed with angiography and/or OCT
Time Frame: During PCI prior to stent implantation (typically 30 min from start of procedure)
Measure: Count of Participants; unit: Participants
Arm/Group | Standalone Percutaneous Coronary Intervention | Percutaneous Coronary Intervention and Thrombus Aspiration | Percutaneous Coronary Intervention and Retriever Thrombectomy
Number analyzed (Participants) | 27 | 27 | 27
Participants | 0 | 0 | 0

3. Primary Outcome: Device Deficiency
Description: Assessed with angiography and/or OCT
Time Frame: During PCI prior to stent implantation (typically 30 min from start of procedure)
Measure: Count of Participants; unit: Participants
Arm/Group | Standalone Percutaneous Coronary Intervention | Percutaneous Coronary Intervention and Thrombus Aspiration | Percutaneous Coronary Intervention and Retriever Thrombectomy
Number analyzed (Participants) | 27 | 27 | 27
Participants | 0 | 0 | 0

4. Primary Outcome: Major Adverse Cardiac and Cerebrovascular Events (MACCE)
Time Frame: Up to 30 days after PCI
Measure: Count of Participants; unit: Participants
Arm/Group | Standalone Percutaneous Coronary Intervention | Percutaneous Coronary Intervention and Thrombus Aspiration | Percutaneous Coronary Intervention and Retriever Thrombectomy
Number analyzed (Participants) | 27 | 27 | 27
Participants | 2 | 4 | 0

5. Primary Outcome: MACCE
Time Frame: At 6 months after PCI
Population: MACCE not available to all participants as two withdrew their consent for participation.
Measure: Count of Participants; unit: Participants
Arm/Group | Standalone Percutaneous Coronary Intervention | Percutaneous Coronary Intervention and Thrombus Aspiration | Percutaneous Coronary Intervention and Retriever Thrombectomy
Number analyzed (Participants) | 26 | 26 | 27
Participants | 5 | 4 | 0

6. Secondary Outcome: Flow Volume (mm^3)
Description: Assessed with OCT
Time Frame: During PCI prior to stent implantation (typically 30 min from start of procedure)
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: mm^3
Arm/Group | Standalone Percutaneous Coronary Intervention | Percutaneous Coronary Intervention and Thrombus Aspiration | Percutaneous Coronary Intervention and Retriever Thrombectomy
Number analyzed (Participants) | 27 | 26 | 27
mm^3 | 30.6 [19.7 to 65.0] | 35.9 [15.1 to 91.7] | 66.5 [41.8 to 108.6]

7. Secondary Outcome: Thromboatheroma Volume (mm^3)
Description: Assessed with OCT
Time Frame: Post-stent implantation during PCI (typically 50 min after procedure start)
Population: One patient was crossed over to direct stent implantation due to radial spasm precluding stent retriever thrombectomy. The OCT runs for some patients were not analysable due to slow flow precluding good blood clearance for a reliable measurement.
Measure: Median (Inter-Quartile Range); unit: mm^3
Arm/Group | Standalone Percutaneous Coronary Intervention | Percutaneous Coronary Intervention and Thrombus Aspiration | Percutaneous Coronary Intervention and Retriever Thrombectomy
Number analyzed (Participants) | 28 | 26 | 24
mm^3 | 3.4 [1.1 to 6.3] | 1.8 [0.6 to 4.7] | 0.5 [0.0 to 2.8]

8. Secondary Outcome: Flow Volume (mm^3)
Description: Assessed with OCT
Time Frame: Post-stent implantation during PCI (typically 50 min after procedure start)
Population: as for outcome 7
Measure: Median (Inter-Quartile Range); unit: mm^3
Arm/Group | Standalone Percutaneous Coronary Intervention | Percutaneous Coronary Intervention and Thrombus Aspiration | Percutaneous Coronary Intervention and Retriever Thrombectomy
Number analyzed (Participants) | 28 | 26 | 24
mm^3 | 5.9 [4.7 to 7.1] | 6.3 [5.0 to 7.4] | 7.2 [5.4 to 8.7]

9. Secondary Outcome: Number of Participants With Stent Underexpansion & Malapposition
Description: Assessed with OCT according to established international consensus criteria.
Time Frame: Post-stent implantation during PCI (typically 50 min after procedure start)
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Standalone Percutaneous Coronary Intervention | Percutaneous Coronary Intervention and Thrombus Aspiration | Percutaneous Coronary Intervention and Retriever Thrombectomy
Number analyzed (Participants) | 28 | 26 | 24
Participants | 5 | 3 | 2

10. Secondary Outcome: Thrombolysis in Myocardial Infarction (TIMI) Flow
Description: Assessed with angiography according to the TIMI Flow criteria
Time Frame: Post-stent implantation during PCI (typically 60 min after procedure start)
Population: TIMI less than 3
Measure: Count of Participants; unit: Participants
Arm/Group | Standalone Percutaneous Coronary Intervention | Percutaneous Coronary Intervention and Thrombus Aspiration | Percutaneous Coronary Intervention and Retriever Thrombectomy
Number analyzed (Participants) | 27 | 27 | 27
Participants | 10 | 5 | 5

11. Secondary Outcome: Number of Participants With Myocardial Blush Grade (MBG) < 3
Description: Assessed angiographically according to the TIMI Myocardial Blush Grade Score Criteria. The scale goes from 0-3. Myocardial blush grade (MGB) of 0, 1 and 2 indicates angiographic malperfusion, whilst a Myocardial blush grade (MGB) score of 3 indicates normal perfusion.
Time Frame: Post-stent implantation during PCI (typically 60 min after procedure start)
Measure: Count of Participants; unit: Participants
Arm/Group | Standalone Percutaneous Coronary Intervention | Percutaneous Coronary Intervention and Thrombus Aspiration | Percutaneous Coronary Intervention and Retriever Thrombectomy
Number analyzed (Participants) | 27 | 27 | 27
Participants | 14 | 6 | 6

12. Secondary Outcome: Angiograpicy Derived Index of Microcirculatory Resistance
Description: The angiography derived index of microcirculatory resistance is a continuous variable that measures microcirculatory resistance. No formal minimum and maximum values exist. The higher the value, the worse the angiographic perfusion. A value over 40U confers an adverse prognosis.
Time Frame: Post-stent implantation during PCI (typically 60 min after procedure start)
Population: The measurement was secondary and to the discretion of the treating physician.
Measure: Median (Inter-Quartile Range); unit: units
Arm/Group | Standalone Percutaneous Coronary Intervention | Percutaneous Coronary Intervention and Thrombus Aspiration | Percutaneous Coronary Intervention and Retriever Thrombectomy
Number analyzed (Participants) | 23 | 22 | 19
units | 50.0 [35.8 to 74.0] | 41 [30.9 to 47.9] | 40.6 [35.7 to 50.1]

ADVERSE EVENTS:
Time Frame: Adverse events were captured at 6 months.
Description: The events recorded in the MACCE section are not adverse events, but rather protocol prespecified clinical endpoints.
Arm/Group | Standalone Percutaneous Coronary Intervention | Percutaneous Coronary Intervention and Thrombus Aspiration | Percutaneous Coronary Intervention and Retriever Thrombectomy
All-Cause Mortality (participants affected / at risk) | 2/27 | 1/27 | 0/27
Serious Adverse Events (participants affected / at risk) | 5/27 | 4/27 | 1/27
Other Adverse Events (participants affected / at risk) | 0/27 | 2/27 | 4/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standalone Percutaneous Coronary Intervention (N=27) | Percutaneous Coronary Intervention and Thrombus Aspiration (N=27) | Percutaneous Coronary Intervention and Retriever Thrombectomy (N=27)
Arrhtymia Related Unplanned Admission (Cardiac disorders) | 1 (1) | 3 (3) | 1 (1) — Arrhythmia requiring admission at 6 months
Death (Prespecified clinical endpoint) (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) — All Cause mortality at 6 months
Chest discomfort (General disorders) | 1 (1) | 0 (0) | 0 (0) — Admission with chest discomfort at 6 months
Major GI Bleeding (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) — Major GI Bleeding Admission
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standalone Percutaneous Coronary Intervention (N=27) | Percutaneous Coronary Intervention and Thrombus Aspiration (N=27) | Percutaneous Coronary Intervention and Retriever Thrombectomy (N=27)
Symptomatic Hypotension (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) — Admission for symptomatic hypotension
Arrhtymia Related Unplanned Admission (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) — Arrhtymia Related Unplanned Admission
Chest discomfort (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2) — Admission of Chest discomfort

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-04-22): https://cdn.clinicaltrials.gov/large-docs/65/NCT05307965/Prot_SAP_000.pdf